CLINICAL TRIAL: NCT05686512
Title: Initial Evaluation of a Stepped Care Model for Treating Mild to Moderate Childhood Anxiety in Primary Care: A Randomized Controlled Feasibility Trial
Brief Title: Initial Evaluation of a Stepped Care Model for Treating Mild to Moderate Childhood Anxiety in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: jaai01
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single-blind parallel-group pilot randomised controlled feasibility trial
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting 12 weeks-assessments will be blind to treatment allocation. The outcome measure (PARS) is identical for both groups, ensuring that the assessors remain blind. At the 12 week-assessment, participants will be reminded to not reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step-by-Step treatment (Experimental): Stepped care cognitive behavioral therapy
  Interventions: Behavioral: Step-by-Step
- Cool Kids treatment (Experimental): Cognitive behavioral therapy
  Interventions: Behavioral: Cool Kids

INTERVENTIONS:
Behavioral: Step-by-Step — The Step-by-Step follows a stepped care approach, were all children (and caregivers) complete the first step (a brief group intervention followed by an individual session). Those with more needs are offered to continue to step 2 where individual CBT is given. See Figure 1 for a schematic representation of the stepped care approach, and Table 2 for an overview of session content.
  Step 1 Session 1-4: Group sessions including psychoeducation, parenting skills and mapping stress and vulnerability factors, exposure and coping skills (90 minutes) Session 5: Individual session - If ending after step 1 a maintenance plan is completed. If continuing to step 2 continued exposure and selection of optional focus areas such as emotion regulation, social skills, stress- and vulnerability factors, child worry or parental worry. (45 minutes)
  Step 2 Session 6-8: Individual sessions - Exposure and selected focus areas. (45 minutes)
  Arms: Step-by-Step treatment
Behavioral: Cool Kids — The Cool Kids Program is an Australian manualized group CBT treatment of child anxiety, which has been broadly implemented in Sweden. Several studies have found evidence of its efficacy.
  Session 1-10: Group sessions including psychoeducation, cognitive restructuring (gather evidence to reevaluate anxiety related thoughts), parent skills, exposure, social skills, coping skills (cognitive and behavioral strategies to handle anxiety reactions, learning problem-solving skills). (120 minutes)
  Arms: Cool Kids treatment

SUMMARY:
Objectives: In the past ten years in Sweden, a new form of primary care units called first line mental health (FLMH) has been implemented to improve mental health services for children and adolescents. Using a structured and collaborative approach including experts, clinicians, and patients, the investigators have developed a transdiagnostic psychological intervention for anxiety based on cognitive behavioural therapy (CBT) that aims to fit the FLMH care context. The current study aims to test the CBT intervention "Step-by-Step" in a randomized pilot study (N=36) to explore the feasibility of the study design.

Rationale for study: Childhood anxiety is common and associated with suffering and impairment in several life areas. CBT is an evidence-based treatment for anxiety disorders in children, but there is a need of increasing access to treatment. Offering CBT for childhood anxiety in primary care is a way to offer early and accessible treatment. However, there is a lack of CBT interventions developed for and evaluated in primary care.

Prior to a properly powered randomized controlled study, evaluating efficacy of the Step-by-Step, the investigators need to conduct a pilot study to, primarily, establish the feasibility of the study design and trial procedures and secondarily, provide preliminary data on acceptability and clinical efficacy.

DETAILED DESCRIPTION:
INTRODUCTION Anxiety is the most common reason for contact with the first line mental health (FLMH) in Sweden. Anxiety disorders are associated with negative effects in several life areas such as school functioning, peer relationships, and family life. Anxiety disorders in children also predict a number of adverse future events such as depression, alcohol and drug abuse, suicide-attempts, and financial problems in young adulthood. Increasing access to evidence-based interventions (EBIs) for child and adolescent anxiety is an urgent task. Today, only a few children and adolescents with life-interfering anxiety use mental health services.

CBT is a treatment that usually involves efforts to change behavioral and thinking patterns. Numerous studies have found evidence for the efficacy of CBT in the treatment of child anxiety, but typically, these treatment programs have been developed for use in a psychiatric setting. The FLMH assignment focuses on early interventions (prevention and treatment) delivered to children and adolescents (and their parents) with mild to moderate mental health problems. A challenge for the FLMH services has been to identify EBIs for anxiety that fit the needs of their patients and their organization, as the available EBIs almost exclusively have been evaluated within the psychiatric domain (i.e., specialist care) rather than with primary care in mind. To solve this problem, FLMH services sometimes offer a full-length EBI, although it does not fit well into the primary care setting (typically the 10 session CBT group program Cool Kids). Or, more commonly, they shorten the intervention despite that empirical support is lacking concerning whether this can be done with maintained treatment efficacy.

Just because an intervention is evidence-based, it does not always fit seamlessly into a certain care setting. The context where the intervention was developed and tested often differ in substantive ways from the context where it is applied. For instance, staff training, resources and patient characteristics might be different. These differences between health care contexts means that EBIs often need to be adapted to fit with the new context. In the FLMH guidelines, CBT is the recommended intervention for child and adolescent anxiety. However, these guidelines refer to studies of comprehensive interventions, typically including ten or more sessions, developed for children with manifest clinical disorders. Consequently, providing CBT within the FLMH means a dilemma concerned with the extent to which the intervention needs to adhere to the original version and the extent to which changes in response to resource restraints and possibilities in the local care context can be done with maintained treatment acceptability and efficacy.

Recently, the investigators have used a structured co-creative approach to develop a CBT intervention to the FLMH in preparation for the current project. The investigators have conducted workshops with experts on CBT for childhood anxiety and with clinicians and heads of three FLMH units. The investigators have also interviewed parents with experience of participating (together with their child) in CBT for childhood anxiety. Based on this information the investigators have developed a treatment called "Step by Step", a stepped care approach to treat anxiety within primary care. During the past months, the investigators have also preliminary tested the acceptability, appropriateness, and feasibility of the Step-by-Step at one FLMH-unit, including 4 participants. Individual qualitative interviews were conducted with therapists, participating children and caregivers after completing the intervention. Interview data was analyzed using thematic analysis.

OBJECTIVES The overarching aim with this research project is to increase the availability to evidence-based psychological treatments for children with anxiety treated within primary care.

Primary Objective: To test the Step-by-Step treatment compared to Cool Kids (an evidence-based treatment) in a randomized pilot study (N=36), to explore the feasibility of the study design.

Secondary Objective: To provide preliminary data on acceptability and clinical efficacy.

PROJECT DESCRIPTION Control group justification: The choice of type of control condition in a trial for a psychological intervention will depend on several factors including the disease and its characteristics, the development phase, the purpose of the study, and the resources available. The investigators decided on Cool Kids for the following reasons: (a) The investigators are interested in comparing Step-by-Step to Cool Kids, to see in a future larger trial if the Step-by-Step is non-inferior to a (comprehensive) evidence-based treatment. (b) The Cool Kids is the most implemented treatment for childhood anxiety in Sweden (both in primary care and in the child- and adolescent psychiatry). (c) Waitlist would not be an ethical choice because there are efficient treatment options available for anxiety in children.

Study Setting: The project will be located at four FLMH-units in Sweden.

Power Analysis: The aim of the study is to evaluate feasibility and acceptability. The investigators have not made any calculation of statistical power, as the investigators do not intend to use inferential statistics in the analyses. There will be 36 participants included, which means three Step-by-Step groups and three Cool Kids groups. The investigators consider this number of children to be suitable to get a broad picture of feasibility and acceptability. The study will be conducted at different FLMH-units, which the investigators consider important to assess the feasibility of our study design.

Data collection: Demographic information (e.g., age, sex, caregivers' educational level, country of birth for caregivers and children) will be collected at baseline and summarized descriptively in sample characteristics. Trial feasibility data (e.g., number of recruited participants, completion rates of the intervention and assessments) will be collected and summarized using descriptive statistics. Clinician-rated anxiety will be administrated by a trained FLMH-therapist at baseline before randomization. At post intervention (defined as 12 weeks after the start of the intervention), the clinician-rated anxiety will be conducted by a trained assessor blinded to treatment allocation. Child-and parent-rated anxiety will be assessed at baseline and 12 weeks after the start of the intervention.

Screening and recruitment procedures: At first visit at the FLMH-unit, the caregiver(s) and the child meet a therapist. The therapist typically collects information about the medical history (including potential previous mental health problems) of the child, assess the severity of mental distress and the global function of the child. If the eligibility criteria are met, the child and caregiver(s) will receive written and verbal information about the study and will be given opportunity to ask questions about the study. If interested in participation, informed written consent will be obtained from all caregivers and the child. If not eligible or interested in participation, patients will be offered regular care at the FLMH-unit (which may include the Cool Kids program or non-manualized individual CBT). If there is a need of contact with specialized psychiatric care and/or other organizations than FLMH (i.e., social services or school) families will be referred according to standard routines at the FLMH units.

Randomization, enrolment and masking: Participants will be randomised at a 1:1 ratio to Step-by-Step or the Cool Kids. Randomisation and masking procedures will be conducted by a researcher in the research group not involved in the clinical aspects of the study. Each FLMH-unit will receive 12 sealed envelopes with six Step-by-Step and six Cool Kids allocations numbered between 1-12. The investigators will use a block-randomization, with block sizes (randomly varying) of 2 and 4. The randomization will be generated using a computer random number generator.

Training and monitoring: All assessors/therapists will receive adequate training before the trial starts. Assessors (i.e., all assessors at the FLMH-units and follow-up assessors) will have received training in the PARS by the doctoral student and psychologist Albin Isaksson. Cool Kids therapists will have received a 2-days training by Skåne certified "train the trainers" at the Skåne child and adolescent psychiatry. Step-by-Step therapists will have received a half day training by psychologists at Gustavsbergs health center (who have experience from running the Step-by-Step in small-scale testing). Adherence to the treatment manuals will be evaluated by independent assessment of a random selection of 25% of the audio recorded sessions. Protocol violations will be recorded.

END OF TRIAL The trial will end when the final data (at the 12-week assessment) has been collected for the final participant. Participants are free to withdraw from the study at any point. After the withdrawal, participants will not be requested to complete any further measures but will be asked to provide non-obligatory feedback regarding their reason for withdrawal. This reason (if given) will be logged for reporting purposes. Withdrawn participants will not be replaced in the trial.

Outcome measures will not be analysed until the end of the trial period and will therefore not inform decisions to stop the research. As the research is conducted within regular first-line operations, professional obligations and the units' routines are followed to handle issues related to patient safety. If during assessment, during an ongoing intervention or in connection with the end of an intervention, a need for care at a different level of care (e.g., in the case of serious psychiatric problems) or a need for interventions from another agency (e.g. due to abuse by a parent) emerges, exposure to violence or neglect) participants will be referred or referred to the appropriate agency.

DATA MANAGEMENT All aspects of data management of the trial will comply with the General Data Protection Regulation and good clinical practice.

Data collection and handling: Audio recordings will be stored on a secure server. Upon inclusion in the pilot study, each participant is assigned an ID number that replaces name and social security number. A code key is established to connect the participant ID and associated data to the participant's personal data. As the study is carried out in a clinical environment, the notes are made in medical records as standard routine. All data collection is monitored by the responsible researcher and PhD student in the project.

BASS: BASS is the name of the data collection tool. BASS is used both for manual entry of clinician assessed/gathered information, as well as for remote (via the internet) administration of child- and parent-reported questionnaires. Regardless of the method above, all data goes into the same database.

ELIGIBILITY:
Inclusion Criteria:

* The child is 7-12 years old. Confirmed by the caregiver and subsequently by the medical records.
* The child suffers from mild to moderate anxiety. The term "mild to moderate anxiety" has not been explicitly defined but is a term aimed to specify a demarcation between the FLMH and the psychiatric specialist services. Adequate level of care for the patient is decided based on an overall clinical assessment. The Children Global Assessment Scale (CGAS) is often used to guide the decision on level of care, where a CGAS value above 60 clearly indicates primary care services, a value below 50 clearly indicates specialist services. For values between 50 and 60 the overall clinical evaluation of symptom severity and impaired function guide the decision on level of care. Confirmed by the assessor at the FLMH-unit

Exclusion Criteria:

* Other psychiatric or developmental disorders than anxiety, or social issues that primarily require other interventions (i.e., where an intervention targeting mild to moderate anxiety is not adequate). Confirmed by assessor at the FLMH-unit.
* The child has another ongoing psychological intervention. An ongoing psychological treatment for any other psychiatric disorder. Confirmed by the caregiver.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment pace | Post intervention (defined as 12 weeks after the start of the intervention)
  Number of included patients per month will be registered for each first line mental health unit, to explore the feasibility of conducting a full scale randomized controlled trial.
Time between first assessment and treatment initiation | Post intervention (defined as 12 weeks after the start of the intervention)
  The investigators will explore number of days between first assessment and treatment initiation to explore if patients do access treatment within a reasonable period of time?
Treatment hours | Post intervention (defined as 12 weeks after the start of the intervention)
  Based on patients' attendance in treatment, therapist time for each patient will be calculated. (For group sessions, hours will be multiplied by number of therapists, and divided by number of patients)
Therapists' views of the intervention | Post intervention (defined as 12 weeks after the start of the intervention)
  A eight item questionnaire will be rated by therapists regarding different aspects of the acceptability, appropriateness, and the feasibility of the intervention content and format.
Patient completion rate | Post intervention (defined as 12 weeks after the start of the intervention)
  Based on patients' attendance in treatment, the investigators will calculate how many patients that attend more than 70% of the sessions.

SECONDARY OUTCOMES:
Treatment credibility inventory (parent- and child-rated) | Two weeks after the start of the treatment
  Four qualitative questions about treatment credibility will be administered after session 2, asking how well the treatment suits children with anxiety, how much they believe this treatment will help him/her, if and to what extent they would recommend this treatment to a friend with depression and how much improvement they expect from the treatment. Each item is scored on a 5-point Likert scale, from 1 to 5. The questionnaire takes around 1 minute to complete.
Client Satisfaction Questionnaire, CSQ (parent-rated) | Post intervention (defined as 12 weeks after the start of the intervention)
  The CSQ is an 8-item self-rated on a 4-point scale measuring different aspects of satisfaction with treatment, e.g., perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction.
Working Alliance Inventory, WAI (parent rated) | Post intervention (defined as 12 weeks after the start of the intervention)
  The WAI is a 6-item scale measuring the participants perceived working alliance with their therapist. The scale is used to control for non-specific therapeutic effects between the different treatment conditions. The questionnaire takes less than 5 minutes to complete.
The Pediatric Anxiety Rating Scale, PARS (clinician rated) | Post intervention (defined as 12 weeks after the start of the intervention)]
  The PARS is a semi-structured clinical interview aimed to assess the severity and functional impairment of anxiety in children aged 6-17 years. Questions are asked to both children and parents. The ratings of severity and impairment is made based on the overall picture of anxiety symptoms. Psychometric evaluations of PARS have shown good psychometric properties of the instrument. PARS has also been used as an outcome measure in several treatment studies.
The Pediatric Anxiety Rating Scale - self-rated, PARS-SR (parent- and child-rated) | Post intervention (defined as 12 weeks after the start of the intervention)
  PARS-SR is a self-rated, brief version of the original clinician-rated PARS that aims to assess the severity of anxiety symptoms associated with common anxiety disorders. The self-rated version has been adapted and translated by our research group, and we have an ongoing study where we will evaluate the psychometric properties in a clinical and school sample.
The Revised Children's Anxiety and Depression Scale-25, RCADS-25 (parent- and child-rated) | Post intervention (defined as 12 weeks after the start of the intervention)
  RCADS-25 is a short version of the original RCADS, developed to measure anxiety symptoms (e.g. "I worry when I think I have done poorly at something") and depressive symptoms (e.g. "I feel sad or empty"). It has two subscales (broad anxiety and depression). All items assess the frequency of symptoms and are rated on a 4-point Likert scale with higher scores indicating more anxiety or depression. The self-report version of RCADS-25 is recommended to use between the ages of 8-18.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Åhlén, PhD, Principal Investigator — Center for epidemiology and community medicine (CES), Stockholm Region
Locations (1):
- Center for epidemiology and community medicine (CES), Stockholm Region, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Only metadata is published openly, underlying data is made available upon request after ensuring compliance with relevant legislation and Region Stockholm guidelines
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Study protocol, ICF will be publicly available at osf.io in February-2023, and Analytic code will be available in (anticipated) November 2023.
Access Criteria: Underlying data is made available upon request after ensuring compliance with relevant legislation and Region Stockholm guidelines